CLINICAL TRIAL: NCT04000152
Title: Randomized Controlled Clinical Study to Assess the Benefit of Non-invasive PGT-A, by the Analysis of Spent Blastocyst Media, as a Tool for Embryo Prioritization in Infertile Patients Undergoing Assisted Reproduction.
Brief Title: RCT Study to Validate niPGT-A Clinical Benefit.
Acronym: niPGT-A_RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment was halted on Mar 1st 2024, after the Data Monitoring Committee, due to low recruitment speed and sustained high dropout rate. Other elements impacted negatively, including the SARS-COV-2 pandemic or the inability to include new sites
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IGX1-NIP-CS-18-05
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Aneuploidy; Chromosome Abnormality; Infertility
Keywords: Blastocyst; Non-invasive; PGT-A; Aneuploidy; Spent culture medium; Trophectoderm biopsy; Sustained implantation; Miscarriage; Livebirth
MeSH Terms: conditions — Aneuploidy; Chromosome Aberrations; Infertility; Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (group 1) (Active Comparator): Deferred single day 6/7 blastocyst transfer with blastocyst selection according to morphology.
  Interventions: Other: Morphology criteria
- Intervention group (group 2) (Experimental): Deferred single day 6/7 blastocyst transfer with blastocyst selection according to the analysis of the spent culture media (niPGT-A).
  Interventions: Diagnostic Test: niPGT-A

INTERVENTIONS:
Diagnostic Test: niPGT-A — Two scenarios should be considered according to the results in the SBM analysis:
  1. The couple decides to transfer the blastocyst selected according to the SBM result (blastocyst prioritization system).
  2. The couple decides to biopsy the blastocysts (if SBM results show low euploidy score). This PGT-A analysis will be offered for free but the outcome of these transfers will be excluded for the analysis per completed protocol. However, all transfers will be included in the intention-to-treat analysis.
  In the exceptional case of getting a non-informative result for all the SBM analysed, the niPGT-A could be performed again on new SBM samples collected after an additional culture of the embryos for, at least, 8 hours.
  Arms: Intervention group (group 2)
Other: Morphology criteria — Embryos for transfer will be selected by the only applicable technique, the assessment of morphology according to Gardner´s criteria, which is the most standardized method.
  Arms: Control group (group 1)

SUMMARY:
Chromosomal aneuploidies are linked with spontaneous miscarriages and abnormal offspring in human pregnancies. In addition, some types of aneuploidies are reported to prevent implantation. Thus, there is a need to identify the embryos with highest implantation potential on in vitro fertilization (IVF) programs.

Since embryo morphology and kinetics have a weak association with embryo ploidy, trophectoderm biopsy plus Next-Generation Sequencing (NGS) is becoming a very popular approach to determine the embryo chromosomal status. This technique is called Preimplantation Genetic Testing for Aneuploidy (PGT-A). Although shown to be efficient, it is invasive for the embryo, requires specific technical skills and it remains expensive. Therefore, the development of a non-invasive, rapid and cheaper method for assessing embryo ploidy status would represent a progress in the field of IVF.

The non-invasive approach has been explored by some groups that analyzed the Spent Blastocyst Medium (SBM) where the embryo was incubated up to the time of transfer or freezing. In daily routine, this media is discarded after finishing the culture of the embryo. Importantly, though, this media reportedly contains traces of embryonic cell-free DNA (cfDNA) that can represent the genetic load of the embryo.

On the basis of that, the hypothesis of this study is that embryo prioritization according to the analysis of the embryonic cfDNA in the SBM could improve ongoing pregnancy rate in 10 percentual points compared to standard blastocyst transfer based on morphology.

DETAILED DESCRIPTION:
Current Preimplantation Genetic Testing for Aneuploidy (PGT-A) techniques analyze the full chromosome content of a single or few cells with high sensitivity and specificity using Next-Generation Sequencing (NGS). Although shown to be efficient, the technique suffers from some limitations. It requires an embryo biopsy, specific technical skills and it still remains expensive. Therefore, non-invasive techniques for assessing embryo ploidy status are sought as an alternative. Such non-invasive approaches would have various advantages over current strategies, including the elimination of a costly micromanipulation biopsy procedure and the avoidance of risks associated with cell removal. Furthermore, it would be more advantageous, especially for those patients who undergo in vitro fertilization (IVF) treatment but do not have PGT-A indication or they are not willing to have their embryos tested with invasive techniques.

One of the recent advances in the field is the identification of embryonic cell-free DNA (cfDNA) during embryo culture in the lab. It is released to the culture drop (SBM) and represents the chromosome content of the embryo. In a recent pilot study, we analyzed the concordance rates between trophectoderm (TE) biopsy and SBM. In SBM collected on day 6/7 of development, the results were concordant with TE biopsies in 84% of samples, with a false-positive rate of 8.6% and a false-negative rate of 2.5%. These findings are encouraging and were the base for the design of the current RCT study.

The main objective of this study is to evaluate the potential clinical benefits of a new non-invasive method for PGT-A, based on the analysis of the embryonic cfDNA released into SBM.

Considering a dropout rate of around 30% (mainly due to treatment or monitoring failures and no day 6/7 blastocysts to transfer), a total of 1108 participants will be randomized before the ovum pick-up. They will be allocated on a balanced way (1:1 ratio) in one of the two arms: 1) Deferred transfer of a single frozen day 6/7 blastocyst which selection was based on the chromosomal status according to the analysis of the SBM; 2) Deferred transfer of a single frozen day 6/7 blastocyst which selection was based on standard embryo morphology (Gardner criteria). Reproductive outcomes (defined following The International Glossary on Infertility and Fertility Care, 2017) will be compared between the two groups.

As this is an open study, both physician and patient will receive the results of the analysis of the culture media. The control group will also have access to these results but at the end of their participation in the study and if she or her physician request it. Additional tests of chromosomal abnormalities (NIPT and POC) could be performed (with no extra cost) under request to ensure patient´s safety and efficacy of the SBM analysis.

Data exported from the medical records and source documents will be duly codified to protect the clinical and personal information of patients in accordance with the current legislation. This information will be exported to an electronic Case Report Form (eCRF). An interim analysis of this data is planned once 30% of the recruitment has been reached. Besides, the study will be overseen by an independent Data Monitoring Committee after 30% of patients´ recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose written informed consent approved by the Ethics Committee (EC) has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
* IVF patients intending to undergo deferred day 6/7 blastocyst SET for any medical indication.
* All the oocytes/embryos from the cycle should follow the laboratory protocol described in the study (embryo culture and vitrification on day 6/7).
* ICSI, IVF or ICSI/IVF performed in fresh own oocytes from couples not undergoing PGT-A. Note: Donor sperm is allowed.
* Female age: 20-40 years, both included.

Exclusion Criteria:

* Assisted hatching and artificial collapse before collecting SBM samples. Note: Both procedures are allowed only after collecting the culture media sample.
* A known abnormal karyotype if the couple provides it at consultation. If not, karyotype is not compulsory.
* Couples planning to undergo PGT-M or PGT-SR cases will be excluded.
* Surrogate pregnancy (in those countries where it is allowed).
* ERA test and embryo transfer according to ERA result.
* Time-lapse culture systems are not allowed after day 4 of culture.
* Presence of pathologies or malformations that affect the uterine cavity such as polyps, intramural myomas ≥ 4cm or submucosal, septum or hydrosalpinx during the patient's participation in the study. Patients suffering these pathologies before or after their inclusion in the study can participate if the pathology is corrected before performing any study procedure.
* Any illness or medical condition that is unstable or which, according to medical criteria, may put at risk the patient's safety and her compliance in the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — IVF patients between 20 and 40 years of age undergoing fertility treatment with their own oocytes, with no intention or medical indication for PGT-A.
Enrollment: 296 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Non-invasive analysis of the chromosomal status of the embryo | 7 days
  Number and structure of the embryo chromosomes
Ongoing pregnancy rate | Over 12 weeks
  Number of ongoing pregnancies per single embryo transfer

SECONDARY OUTCOMES:
NGS results of the SBM | 7 days at least
  Informativity rates and prioritization category of the SBM analysis results with embryo development, culture conditions and collection time
Non-Invasive Prenatal Testing (NIPT) | Up to 12 weeks
  Incidence of chromosomal abnormalities in NIPT within ongoing pregnancy cases
Clinical miscarriage rate | Up to 6 months after the ovum pick-up
  Number of clinical miscarriages per total number of ongoing pregnancies
Analysis of the Products of Conception (POC) | Up to 20 weeks
  Incidence of chromosomal abnormalities in POC within miscarriage cases
Cumulative ongoing pregnancy rate | Over 6 months after the ovum pick-up
  Cumulative ongoing pregnancy rate per patient in the 6 months after the pick-up
Time to get an ongoing pregnancy | Up to 6 months after the ovum pick-up
  Time to get an ongoing pregnancy within the 6 months after the pick-up
Live birth rate | Over 40 weeks
  Number of babies born per embryo transfer
Cumulative live birth rate | Over 6 months after the ovum pick-up
  Cumulative live birth rate per patient in the 6 months after the pick-up
Obstetrical outcomes comparison | Over 40 weeks
  To compare birth weight, gestational age, APGAR, type of delivery, pregnancy complications, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Rubio, PhD, Principal Investigator — Igenomix S.L.
Locations (8):
- Argentina (2):
  - Crecer: Centro de Reproducción y Genética Humana, Mar del Plata, Buenos Aires
  - Saresa - Reproducción Humana Asistida, Salta, Salta Province
- Brazil (2):
  - Nilo Frantz - Centro de Reprodução Humana, Boa Vista, Porto Alegre
  - Vida - Centro de Fertilidade, Rio de Janeiro, Rio de Janeiro
- Hôpital Foch, Suresnes, Suresnes, France
- Italy (2):
  - Società Italiana Studi di Medicina della Riproduzione (S.I.S.M.e.R.), Bologna, Bologna
  - Centro Procreazione Assistita DEMETRA, Florence, Firenze
- Hospital Ruber Internacional, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No